CLINICAL TRIAL: NCT01260519
Title: Efficacy of a Single Dose Intravenous Heparin During Diagnostic Angiography in Reducing Sheath-clot Formation: A Randomized Controlled Trial
Brief Title: Effect of Heparin on Femoral Arterial Sheaths Thrombosis During Diagnostic Coronary Angiography
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prince Sultan Cardiac Center, Adult Cardiology Department. (Other)
Responsible Party: Abdulrahman M Al-Moghairi,MD,MRCP, SFC, Prince Sultan Cardiac Center, Adult Cardiology Department.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PSCC-00001- HT
Record Dates: First submitted 2010-11-19; First posted 2010-12-15 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-12

CONDITIONS: Diagnostic Coronary Angiography
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- active arm: heparin (Experimental)
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Heparin — unfractionated heparin 2000 unites
  Other Names: unfractionated heparin

SUMMARY:
The project tests the incidence of femoral arterial sheath thrombus formation during diagnostic coronary angiography and effect of intravenous (iv) heparin bolus administration in reducing this risk in comparison to placebo.

DETAILED DESCRIPTION:
PURPOSE:

The purpose of this study was to evaluate the incidence of blood clots in femoral arterial sheaths during coronary angiographic procedures and the effect of heparin administration on thrombus formation.

BACKGROUND:

A heparinized saline flushes are used during diagnostic coronary angiography to prevent thrombus formation within the lumen of the sheath. However, the use of prophylactic intravenous heparin following the femoral arterial sheath insertion is controversial. The aim of this study was to evaluate the effectiveness of 2000 units heparin intravenous bolus versus saline placebo on thrombus formation within arterial sheath during the diagnostic coronary angiography.

Methods A randomized controlled trial to examine the efficacy of intravenous heparin bolus compared with placebo in prevention of femoral arterial sheath thrombus formation in patients undergoing diagnostic coronary angiography.

The study included all adult patients undergoing cardiac catheterization. Eligible patients were recruited from day-case and in-patients wards of the Prince Sultan Cardiac Centre (PSCC), Riyadh. Patients with abnormal coagulation profile, abnormal platelet count and those receiving enoxaparin, or glycoprotein IIb/IIa antagonists were excluded.

Since the coronary interventions require anticoagulation during the procedure, our study was interested in the diagnostic part. After insertion of femoral arterial sheath one group was allocated to 2 milliliter solution containing 2000 units of heparin and the other group to similar amount of placebo solution which is blinded to both patient and operating catheterization laboratory staff. Arterial access was obtained via femoral approach and 6F to 7F Sheaths were used. The femoral sheath was aspirated and flushed for presence of thrombi or obstruction after each catheter exchange and at the end of the procedure. Two steps aspiration was performed where 5 cc of blood were extracted in one syringe then another saline filled syringe was used for flushing. We used clean white gauze to look for presence of thrombi, and if thrombi were noticed further aspiration was performed followed by saline flush. Any visible thrombus at any stage of the procedure was considered positive. The patients evaluated and assessed clinically during hospital stay for presence of leg ischemia, Femoral and Pedal pulses, Local hematoma or bleeding.

All patients gave informed consent, and the study protocol was approved by the PSCC Ethics Committee.

Randomization Patients were randomized based catheterization laboratory flow, where the first laboratory assigned to treatment number one and the second laboratory assigned to treatment number two on alternate days, sealed and labeled syringes that contained the treatment allocation came from pharmacy on daily basis and handled to an independent laboratory staff nurse assigned to maintain concealed to patients and healthcare providers Throughout the study. The labels were uncovered opened only after the femoral puncture and arterial sheath insertion confirmed and the patient had provided written informed consent to participate in the study. Once the seal was broken, the patient was considered irrevocably randomized.

Study Interventions Patients were randomized to receive either heparin or placebo. Patients in the heparin group received 2000 units (2 ml) of unfractionated heparin intravenous bolus. Those randomized to the placebo received 2ml of saline based solution intravenous bolus.

The femoral sheath was aspirated and flushed for presence of thrombi or obstruction after each catheter exchange and at the end of the procedure. Two steps aspiration was performed where 5 cc of blood were extracted in one syringe then another saline filled syringe was used for flushing. We used clean white gauze to look for presence of thrombi, and if thrombi were noticed further aspiration was performed followed by saline flush. Any visible thrombus at any stage of the procedure was considered positive. The patients evaluated and assessed clinically during hospital stay for presence of leg ischemia, Femoral and Pedal pulses, Local hematoma or bleeding.

Outcomes The primary end point was the occurrence of arterial sheath thrombi, defined as Any visible thrombus during sheath blood aspiration at any stage of the procedure. The second primary end point was efficacy of intravenous heparin bolus in reducing the risk of thrombus formation.

Patients were monitored for embolic and bleeding events until they were discharged from the hospital. Embolic events defined as appearance of symptoms and signs of acute limb ischemia like acute leg pain and loss of pedal pulses that result in interventional or surgical exploration. Bleeding events was defined as local femoral access bleeding or hematoma that led to surgical exploration.

The diagnosis of embolization or hematoma was made clinically (loss of arterial pulse or evidence of leg ischemia) and confirmed by Doppler studies when appropriate.

Outcomes were assessed by the patients' treating physicians, who were aware of treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

* Included all adult patients undergoing cardiac catheterization

Exclusion Criteria:

* Contraindication to heparin
* Platelet count <100,000/mm3
* Patient with bleeding diathesis or hypercoagulable state.
* Use of chronic anticoagulation with INR > 1.4
* Patient refusal or inability to follow the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2008-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The incidence of femoral arterial sheath thrombi and the efficacy of heparin bolus in preventing sheath thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Abdulrahman M Almoghairi, MD, Principal Investigator — Prince Sultan Cardiac Centre (PSCC)
Locations (1):
- Prince Sultan Cardiac Center, Riyadh, Central, Saudi Arabia